CLINICAL TRIAL: NCT03598075
Title: Amylin and CGRP Migraine Provocation in Migraine Without Aura Patients
Brief Title: Amylin and CGRP Head to Head Provocation in Migraine Without Aura Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, MD, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H-17035931
Record Dates: First submitted 2018-06-28; First posted 2018-07-26 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Islet Amyloid Polypeptide; pramlintide

STUDY DESIGN:
Intervention Model Description: In a Randomized, double blind, cross over experiment. Migraine without aura patients will received amylin or CGRP in two separate days apart by a week.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amylin (Pramlintide) (Other): Pramlintide intravenous infusion 120 micrograms over 20 minutes
  Interventions: Other: Amylin (Pramlintide)
- CGRP (Other): CGRP intravenous infusion 30 micrograms over 20 minutes
  Interventions: Other: CGRP

INTERVENTIONS:
Other: Amylin (Pramlintide) — Pramlintide is a amylin analog. It will be given intravenously at the rate of 120 micrograms over 20 minutes .
  Arms: Amylin (Pramlintide)
Other: CGRP — CGRP It will be given intravenously at the rate of 30 microgram over 20 minutes.
  Arms: CGRP

SUMMARY:
Amylin and calcitonin gene related peptide (CGRP) are related to the same peptide family. Both share 16 out of 37 amino acids and can activate each others receptor. CGRP is implicated in migraine pathophysiology but the role of Amylin and its receptor in migraine is not fully clarified.

DETAILED DESCRIPTION:
Amylin is a peptide hormone that binds to a G-protein coupled receptor (GPCR). amylin was originally found in the pancreas (Beta Cell of Islets of Langerhans) but also shown to be present in the trigeminal ganglion, hind horn ganglia and perivascular nerve fibers.

Amylin has many similarities with CGRP. Amylin and CGRP share 16 out 37 amino acids. Both peptides can activate the amylin 1 subtype (AMY1)receptor with high affinity and reported to have more similar physiological and pharmacological effects.

In addition, both peptides increase the intracellular concentration of cyclic AMP (cAMP) which has a central role in migraine pathophysiology.

The aim of the study is pin point the role of amylin and amylin receptor compare to CGRP in migraine pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients meeting International Headache Society (IHS) criteria for migraine without aura of both sexes, 18-60 year, 50-100 kg.
* Fertile women should use safe contraception. Fertile women do not include hysterectomized women or women who are postmenopausal for at least 2 years. Safe contraception includes either Intra Uterine Device (IUD), birth control pills, surgical sterilization of the woman or depot progestogen.

Exclusion Criteria:

* Tension Type headache for more than 5 days the month on average in the last year.
* All other primary headaches .
* Headache later than 48 hours before trial start.
* Daily intake of any medicine other than oral contraception.
* Ingestion of any form of medicinal product later than 4 times the plasma half-life substance (on trial day), except for oral contraception.
* Pregnant or breastfeeding women.
* Headache on the test day or later than 48 hours prior to administration of trial medicine / placebo
* Migraine within 5 days before the trial date.
* Ancestral information or clinical signs of (on the day of inclusion):
* Hypertension (systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 100 mmHg)
* Hypotension (systolic blood pressure <90 mm Hg and / or diastolic blood pressure <50 mmHg)
* Cardiovascular disease of all kinds, including cerebrovascular disease.
* Anamnestic or clinical signs of mental illness or abuse.
* Patients with glaucoma or prostatic hyperplasia
* Anamnestic or clinical signs of diseases of any kind such as the investigating physician is considered relevant for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Migraine incidence | 12 hours
  Before (-10 min) and after infusion (+12 hours) of amlyin compared with before and after infusion of CGRP based on questionnaire reported headache and associated symptoms

SECONDARY OUTCOMES:
Dilatation of Arteria radialis and arteria temporalis superficialis | 2 hours
  Dermascan will be used to measure the above mentioned Radial and temporal arteries diameter.
Facial flushing | 2 hours
  Flushing will measured by laser contrast imaging
Plasma blood samples | 2 hours
  Measumrent of amylin and CGRP peptides in the plasma in picomol/L
Headache intensity | 12 hours
  Measured by visual analog score (VAS) ( 0 to 10). Change in area under curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No